CLINICAL TRIAL: NCT02194309
Title: Safety, Tolerability and Pharmacokinetics of Single and Multiple Oral Doses of 40 mg Telmisartan/5 mg Amlodipine and 80 mg Telmisartan/5 mg Amlodipine (Free Dose Combination) in Healthy Male Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics of Single and Multiple Oral Doses of 40 mg Telmisartan/5 mg Amlodipine and 80 mg Telmisartan/5 mg Amlodipine in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1235.9
Record Dates: First submitted 2014-07-17; First posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Amlodipine

ARMS (2):
- Telmisartan low + amlodipine (Experimental)
  Interventions: Drug: Telmisartan low; Drug: amlodipine
- Telmisartan high + amlodipine (Experimental)
  Interventions: Drug: Telmisartan high; Drug: amlodipine

INTERVENTIONS:
Drug: Telmisartan low
  Arms: Telmisartan low + amlodipine
Drug: Telmisartan high
  Arms: Telmisartan high + amlodipine
Drug: amlodipine

SUMMARY:
To investigate safety, tolerability, and pharmacokinetics of telmisartan and amlodipine following single administration of 40 mg telmisartan/5 mg amlodipine and 80 mg telmisartan/5 mg amlodipine, and subsequently, following multiple administration of 40 mg telmisartan/5 mg amlodipine and 80 mg telmisartan/5 mg amlodipine once daily for 10 days

ELIGIBILITY:
Inclusion Criteria:

Healthy male volunteers according to the following criteria:

1. No finding deviating of clinical relevance and no evidence of a clinically relevant concomitant disease based upon a complete medical history, including the physical examination, vital signs (blood pressure, pulse rate, body temperature), 12-lead ECG, clinical laboratory tests
2. Age ≥20 and Age ≤35 years
3. Body weight ≥50 kg
4. Body mass index (BMI) ≥17.6 and BMI ≤26.4 kg/m2
5. Signed and dated written informed consent before admission to the trial

Exclusion Criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
3. Chronic or relevant acute infections
4. Any clinical relevant findings of the laboratory test deviating from normal
5. Positive result for either hepatitis B surface antigen (HBsAg), anti hepatitis C virus (HCV) antibodies, syphilitic test or human immunodeficiency virus (HIV) test
6. History of surgery of gastrointestinal tract (except appendectomy)
7. History of relevant orthostatic hypotension (mean standing systolic blood pressure (SBP) varied by ≥20 mmHg from mean supine SBP or mean standing diastolic blood pressure (DBP) varied by ≥10 mmHg from mean supine DBP), fainting spells or blackouts
8. History of hepatic dysfunction (e.g., biliary cirrhosis, cholestasis)
9. History of serious renal dysfunction
10. History of bilateral renal artery stenosis or renal artery stenosis in a solitary kidney
11. History of cerebrovascular disorder
12. History of hyperkalemia
13. Known hypersensitivity to any component of the formulation, or to any other Angiotensin Receptor Blocker (ARB), angiotensin converting enzyme or dihydropyridine
14. Intake of drugs with a long half-life (≥24 hours) within at least one month or less than 10 half-lives of the respective drug before administration or during the trial
15. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 7 days before administration or during the trial
16. Participation in another trial with an investigational drug within 4 months or 6 half-lives of the investigational drug before administration
17. Smoker (≥20 cigarettes/day)
18. Alcohol abuse (60 g or more ethanol/day: ex. 3 middle-sized bottles of beer, 3 gous (equivalent to 540 mL) of sake)
19. Drug abuse
20. Blood donation (more than 100 mL within 4 weeks before administration or during the trial)
21. Excessive physical activities (within 1 week before administration or during the trial)
22. Intake of alcohol within 2 days before administration
23. Inability to comply with dietary regimen of trial centre
24. Intake of any drugs/supplements with ingredient of hypericum perforatum (citrus fruits, Sevilla orange) within 5 days prior to administration
25. Inability to refrain from smoking on trial days

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2006-09; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with clinically significant changes in vital signs (blood pressure, pulse rate, body temperature) | up to 6 days after last administration in multiple dose phase
Number of patients with clinically significant changes in 12-lead electrocardiogram (ECG) | up to 6 days after last administration in multiple dose phase
Number of patients with clinically significant changes in laboratory parameters | up to 6 days after last administration in multiple dose phase
Number of patients with adverse events | up to 6 days after last administration in multiple dose phase
Assessment of tolerability by investigator on a four-point scale | up to 6 days after last administration in multiple dose phase

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) for several time points | up to day 16
tmax (time from dosing to the maximum measured concentration of the analyte in plasma) for several time points | up to day 16
Cmin,ss (minimum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | up to day 16
AUC (area under the concentration-time curve of the analyte in plasma) for several time points | up to day 16
λz (terminal rate constant in plasma) for several time points | up to day 16
t1/2 (terminal half-life of the analyte in plasma) for several time points | up to day 16
MRTpo (mean residence time of the analyte in the body after oral administration) for several time points | up to day 16
CL/F (apparent clearance of the analyte in plasma following extravascular administration) for several time points | up to day 16
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular administration) for several time points | up to day 16
Accumulation ratio (RA) based on Cmax | up to day 16
RA based on AUC | up to day 16
Predose concentration (Cpre) for several time points | up to day 10
C24,10 | 24 hours after last administration on day 10